CLINICAL TRIAL: NCT00433420
Title: A Phase III Randomized Study of EC Followed by Paclitaxel Versus FEC Followed by Paclitaxel, All Given Either Every 3 Weeks or 2 Weeks Supported by Pegfilgrastim, for Node Positive Breast Cancer Patients
Brief Title: Combination Chemotherapy With or Without Fluorouracil and/or Pegfilgrastim in Treating Women With Node-Positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Collaborators: Gruppo Italiano Mammella (GIM) (Other)
Responsible Party: Principal Investigator, Lucia Del Mastro,MD, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Allocation: Randomized | Purpose: Treatment
Other Study IDs: GIM-2; CDR0000528056 (Registry Identifier: PDQ (Physician Data Query)); EU-20681
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pegfilgrastim; Cyclophosphamide; Epirubicin; Fluorouracil; Paclitaxel; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: pegfilgrastim
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: paclitaxel
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epirubicin, cyclophosphamide, paclitaxel, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Colony-stimulating factors, such as pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Giving combination chemotherapy and pegfilgrastim after surgery may kill any tumor cells that remain after surgery. It is not yet known whether combination chemotherapy is more effective with or without fluorouracil and/or pegfilgrastim in treating breast cancer.

PURPOSE: This randomized phase III trial is studying combination chemotherapy to compare how well it works when given with or without fluorouracil and/or pegfilgrastim in treating women with node-positive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of adjuvant therapy comprising epirubicin hydrochloride, cyclophosphamide, and paclitaxel with vs without fluorouracil and/or pegfilgrastim in women with node-positive breast cancer.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Compare the safety of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive epirubicin hydrochloride IV and cyclophosphamide IV on day 1. Treatment repeats every 3 weeks for 4 courses. Patients then receive paclitaxel IV over 3 hours on day 1. Treatment with paclitaxel repeats every 3 weeks for 4 courses.
* Arm II: Patients receive fluorouracil IV, epirubicin hydrochloride IV, and cyclophosphamide IV on day 1. Treatment repeats every 3 weeks for 4 courses. Patients then receive paclitaxel as in arm I.
* Arm III: Patients receive epirubicin hydrochloride IV and cyclophosphamide IV on day 1 and pegfilgrastim subcutaneously (SC) on day 4. Treatment repeats every 2 weeks for 4 courses. Patients then receive paclitaxel IV over 3 hours on day 1 and pegfilgrastim subcutaneously (SC) on day 4. Treatment with paclitaxel and pegfilgrastim repeats every 2 weeks for 4 courses.
* Arm IV: Patients receive fluorouracil IV, epirubicin hydrochloride IV, and cyclophosphamide IV on day 1 and pegfilgrastim SC on day 4. Treatment repeats every 2 weeks for 4 courses. Patients then receive paclitaxel and pegfilgrastim as in arm III.

In all arms, treatment continues in the absence of disease progression or unacceptable toxicity. After completion of chemotherapy with or without pegfilgrastim, patients may undergo external-beam radiation therapy at the discretion of treating center. Patients with positive estrogen and/or progesterone receptor tumor receive tamoxifen for 5 years.

After completion of study treatment, patients are followed periodically for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 2,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary breast cancer

  * No histology other than carcinoma
* Node-positive disease

  * Must have at least 1 involved axillary node or internal mammary node
* Previously resected disease

  * Has undergone radical surgery (i.e., mastectomy or conservative surgery) with axillary node dissection within the past 7 weeks
* No inflammatory carcinoma
* No prior or concurrent ipsilateral or contralateral invasive breast carcinoma
* No metastatic disease, including metastasis in the ipsilateral supraclavicular lymph nodes
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* ECOG performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* WBC ≥ 4,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No chronic liver or renal disease
* No other serious medical illness requiring medication
* No other malignancy except adequately treated, cone-biopsied in situ carcinoma of the cervix or basal cell or squamous cell carcinoma of the skin
* No symptomatic peripheral neuropathy > grade 2
* No hypersensitivity to study drugs or their components
* No recent myocardial infarction, congestive heart failure, or serious arrhythmia

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy
* No prior cytotoxic regimens
* No prior radiation therapy, except for intraoperative radiation therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2003-04 (Actual); Primary Completion 2006-05 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival

SECONDARY OUTCOMES:
Overall survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Marco Venturini, MD, Study Chair — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy

REFERENCES:
- [Derived] Del Mastro L, Poggio F, Blondeaux E, De Placido S, Giuliano M, Forestieri V, De Laurentiis M, Gravina A, Bisagni G, Rimanti A, Turletti A, Nistico C, Vaccaro A, Cognetti F, Fabi A, Gasparro S, Garrone O, Alicicco MG, Urracci Y, Mansutti M, Poletti P, Correale P, Bighin C, Puglisi F, Montemurro F, Colantuoni G, Lambertini M, Boni L; Gruppo Italiano Mammella Investigators. Fluorouracil and dose-dense adjuvant chemotherapy in patients with early-stage breast cancer (GIM2): end-of-study results from a randomised, phase 3 trial. Lancet Oncol. 2022 Dec;23(12):1571-1582. doi: 10.1016/S1470-2045(22)00632-5. Epub 2022 Nov 10. PMID 36370716
- [Derived] Lambertini M, Bruzzi P, Poggio F, Pastorino S, Gardin G, Clavarezza M, Bighin C, Pronzato P, Del Mastro L. Pegfilgrastim administration after 24 or 72 or 96 h to allow dose-dense anthracycline- and taxane-based chemotherapy in breast cancer patients: a single-center experience within the GIM2 randomized phase III trial. Support Care Cancer. 2016 Mar;24(3):1285-94. doi: 10.1007/s00520-015-2907-2. Epub 2015 Aug 27. PMID 26306520
- [Derived] Del Mastro L, De Placido S, Bruzzi P, De Laurentiis M, Boni C, Cavazzini G, Durando A, Turletti A, Nistico C, Valle E, Garrone O, Puglisi F, Montemurro F, Barni S, Ardizzoni A, Gamucci T, Colantuoni G, Giuliano M, Gravina A, Papaldo P, Bighin C, Bisagni G, Forestieri V, Cognetti F; Gruppo Italiano Mammella (GIM) investigators. Fluorouracil and dose-dense chemotherapy in adjuvant treatment of patients with early-stage breast cancer: an open-label, 2 x 2 factorial, randomised phase 3 trial. Lancet. 2015 May 9;385(9980):1863-72. doi: 10.1016/S0140-6736(14)62048-1. Epub 2015 Mar 2. PMID 25740286